CLINICAL TRIAL: NCT01200433
Title: The Effects of Dexmedetomidine and Propofol on Cerebral Blood Flow and Brain Oxygenation During Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ehab Farag, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 10-715
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Intracranial Neurosurgery
Keywords: dexmedetomidine; propofol; cerebral blood flow; brain oxygenation
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol (Active Comparator): Subjects will be sedated with propofol.
  Interventions: Drug: propofol
- dexmedetomidine (Active Comparator): Subjects will be sedated with dexmedetomidine.
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — Patients assigned to dexmedetomidine will be given a mg/kg bolus over 10-20 minutes; subsequently, an infusion will be titrated to between 0.4-0.6 mcg/kg/hr to maintain an adequate level of sedation during the procedure.
  Other Names: Precedex
  Arms: dexmedetomidine
Drug: propofol — Patients assigned to propofol will be given an infusion dose of 50-75 µ/kg/min which will be titrated to the patient's response
  Arms: propofol

SUMMARY:
The investigators will evaluate the effects of dexmedetomidine and propofol on cerebral blood flow and brain oxygenation during Deep Brain Stimulation (DBS) surgery. Specifically, the investigators will test the hypothesis that dexmedetomidine is non-inferior to propofol for cerebral blood flow as measured by transcranial Doppler and brain oxygenation as measured by near-infrared spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III.
* Scheduled for DBS.

Exclusion Criteria:

* History of dystonia.
* Severe heart failure with ejection fraction less than 30%.
* History of obstructive sleep apnea.
* History of renal failure with creatinine level > 2 mg/dl.
* Allergies to α-2 agonists and propofol.
* Current use of α-2 agonist medications such as clonidine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Farag, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farag E, Kot M, Podolyak A, Argalious M, Deogaonkar M, Mascha EJ, Xu Z, Katzan I, Ebrahim Z. The relative effects of dexmedetomidine and propofol on cerebral blood flow velocity and regional brain oxygenation: A randomised noninferiority trial. Eur J Anaesthesiol. 2017 Nov;34(11):732-739. doi: 10.1097/EJA.0000000000000662. PMID 28891839

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol | Dexmedetomidine
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Dexmedetomidine | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.5) | 65.4 (6.8) | 64.5 (8.7)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 18 | 18 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 21 | 21 | 42
  Others | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Blood Flow
Description: Cerebral blood flow was the average of right and left carotid velocities recorded by transcranial Doppler.
Time Frame: For patients randomized to dexmedetomidine: at the first peak of study drug (i.e., at peak dose of study drug during first infusion period); for patients randomized to propofol: when infusion of propofol stopped.
Measure: Median (Inter-Quartile Range); unit: cm/sec
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 21 | 23
cm/sec | 45.4 [37.0 to 48.0] | 39.9 [31.5 to 47.0]
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Non-Inferiority or Equivalence — We tested a joint hypothesis that dexmedetomidine was noninferior to propofol both in terms of cerebral blood flow velocity and brain oxygenation during DBS surgery. A total of 44 patients provided a 90% power at the 0.05 significance level to detect noninferiority of dexmedetomidine to propofol using a noninferiority ratio of geometric means of 0.80, assuming a coefficient of variation of 25% for each of the 2 primary outcomes. Both outcomes were expected to follow a log-normal distribution; p = 0.011, t-test, 1 sided; Ratio of Geometric Means = 0.94, 90% CI 2-sided [0.84 to 1.05] — Dexmedetomidine vs. propofol

2. Primary Outcome: Brain Oxygen
Description: Brain oxygenation values were estimated by near-infrared spectroscopy and brain oxygenation was averaged across the first and second study drug infusion periods.
Time Frame: during first (10-20 minutes) and second (throughout the procedure) study drug infusion periods
Measure: Median (Inter-Quartile Range); unit: % oxygenation
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 21 | 23
% oxygenation | 73.5 [70.3 to 76.6] | 72.7 [70.0 to 75.3]
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 1 sided; Ratio of Geometric Means = 0.99, 90% CI 2-sided [0.96 to 1.02] — Dexmedetomidine vs. propofol

3. Secondary Outcome: Cerebral Blood Flow
Description: The investigator will test the hypothesis that dexmedetomidine is non-inferior to propofol for cerebral blood flow as measured by transcranial Doppler and brain oxygenation as measured by near-infrared spectroscopy.
Time Frame: after procedure, in post anesthesia care unit (PACU)
Population: The cerebral flow at PACU was not planned as a primary outcome. The primary outcome was cerebral flow at the first peak of study drug. The data was collect for information purpose only. No test was done for cerebral blood flow at PACU.
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 21 | 23
cm/sec | 55 (18.1) | 46.7 (10.5)

4. Secondary Outcome: Alertness/Sedation
Description: Modified observer's assessment of alertness /sedation (OAA/S) scale which ranges from 0 to 5 (0 = does not respond to noxious stimuli and 5 = responds to name spoken in normal tone)
Time Frame: at the first peak during DBS surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 21 | 23
units on a scale | 2 [1 to 2] | 3 [2 to 3]
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1, 99% CI 2-sided [0 to 2]

5. Secondary Outcome: Pulsatility Index
Description: Pulsatility index is a measure of the variability of blood velocity in a vessel, and was calculated as the difference between the peak systolic and minimum diastolic velocities divided by the mean velocity during the cardiac cycle.
Time Frame: at the first peak during DBS surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 21 | 23
units on a scale | 1 [0.89 to 1.05] | 1 [0.92 to 1.15]
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Superiority or Other; p = 0.91, Wilcoxon (Mann-Whitney); Ratio of Geometric Means = 1, 99% CI 2-sided [0.86 to 1.18]

6. Secondary Outcome: Cerebral Perfusion Pressure
Time Frame: at the first peak during DBS surgery
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 21 | 23
mmHg | 53.9 [45.1 to 69.8] | 54.6 [48.9 to 66.0]

7. Secondary Outcome: Number of Hypertensive Episodes
Description: The number of hypertensive episodes during Deep Brain Stimulation (DBS) surgery.
Time Frame: During DBS surgery
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 21 | 23
number of episodes | 4.9 (2.7) | 2.9 (2.5)
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.9, 99% CI 2-sided [-4.1 to 0.2]

8. Secondary Outcome: Number of Apneic Episodes.
Description: The number of antihypertensive interventions during Deep Brain Stimulation (DBS) surgery.
Time Frame: during DBS surgery
Measure: Median (Inter-Quartile Range); unit: number of episodes
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 21 | 23
number of episodes | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Propofol vs Dexmedetomidine; Test type: Superiority or Other; p > 0.99, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 99% CI 2-sided [0 to 0]

ADVERSE EVENTS:
Arm/Group | Propofol | Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes